CLINICAL TRIAL: NCT04567069
Title: Phase I/II Study of DC Vaccine Targeting MG-7 Antigen to Treat Gastric Cancer
Brief Title: Safety and Efficacy Study for MG-7-DC Vaccine in Gastric Cancer Treatment
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Shandong University (Other)
Collaborators: Shandong Sunstem Biotechnology Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC-S-Ⅰ/Ⅱ
Record Dates: First submitted 2020-09-23; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, DC vaccine, CTL, MG-7 antigen, PD-1 monoclonal antibody
MeSH Terms: conditions — Stomach Neoplasms | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DC vaccine (Experimental): Vaccine made from autologous dendritic cells loaded with MG-7 antigen.
  Interventions: Biological: DC vaccine
- DC vaccine + CTL (cytotoxic lymphocyte) (Experimental): Cytotoxic lymphocytes are CD3+ T cells co-cultured with DCs.
  Interventions: Biological: DC vaccine; Biological: CTL
- DC vaccine + PD-1 monoclonal antibody (Sintilimab Injection) (Experimental): Sintilimab injection is a type of immunoglobulin G4 monoclonal antibody, which binds to PD-1 molecules on the surface of T-cells, blocks the PD-1/ PD-1 Ligand-1 (PD-L1) pathway and reactivates T-cells to kill cancer cells.
  Interventions: Biological: DC vaccine; Drug: Sintilimab Injection

INTERVENTIONS:
Biological: DC vaccine — Blood samples will be collected twice, 60-120ml/ time. The 1st collection will occur 5 days before the 1st DC vaccine injection, the 2nd collection will occur 15 days after the 1st injection.
  Six subcutaneous(ih) injections of DC vaccine will be given at days 1, 8, 15, 21, 28, 35; 1-3×106 cells/time.
  Injection site: inguinal lymph nodes.
  Other Names: MG-7-DC vaccine; MG-7 antigen-pulsed autologous DC vaccine
Biological: CTL — Four intravenous (iv) drip injections of CTL will be given at days 7, 9, 27, 29; 1-2×109 cells/time.
  Arms: DC vaccine + CTL (cytotoxic lymphocyte)
Drug: Sintilimab Injection — The Sintilimab Injection (3mg/kg) will be administered by intravenous (iv) drip injection at days 0, 20。
  Other Names: Sintilimab; Tyvyt
  Arms: DC vaccine + PD-1 monoclonal antibody (Sintilimab Injection)

SUMMARY:
The primary purpose of the study is to determine the safety and efficacy of autologous DC vaccine in patients with later stage of gastric cancer. The DC vaccine is gene modified with gastric cancer specific antigen MG-7.

DETAILED DESCRIPTION:
All eligible patients will receive two cycles of treatment, every 21 days is a treatment cycle. The follow-up time will start from the next day after the end of the second cycle of treatment, and last for 48 ±1 weeks (the follow-up time is 4 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks). During the treatment and follow-up period, if disease progression or intolerable side effects develop, the patient can voluntarily request to be withdrawn from the study, or the investigators can determine that the patient be removed from the study.

DC and CTL are immune cells. PD-1 monoclonal antibody is an immune checkpoint inhibitor. According to the relevant experience of similar cells or drugs, some patients may have delayed or early pseudo-tumor progression after receiving immunotherapy, which needs to be judged by investigators.

In this study, the screening period is no more than 14 days. After the screening examination and evaluation, the eligible patients will enter the treatment period. The treatment and follow-up are carried out according to the procedure. The follow-up period: tumor imaging evaluation and related clinical indicator evaluation are carried out at the 4th week (± 1 week), the 12th week (± 1 week), the 24th week (± 1 week), the 36th week (± 1 week) and the 48th week (± 1 week) after the treatment. The patients should also complete the corresponding safety inspection and evaluation before leaving the group. During the follow-up period, the patients who do not have disease progression but do leave the group should continue to be evaluated according to the original frequency until the end of the follow-up period or the start of other anti-tumor treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed gastric adenocarcinoma.
2. Patients should be within age range of ≥18 and ≤80 years old, competent, have signed informed consent and have a life expectancy greater than 6 months.
3. Failed in previous standard therapy ( surgery, chemotherapy, radiotherapy, and targeted therapy) or recurred from previous therapy, patients must be at least 1 month from their last therapy.
4. Patients without indications of surgery, radiotherapy or chemotherapy.
5. Patients who can't tolerate radiotherapy or chemotherapy.
6. Patients who refuse radiotherapy or chemotherapy.
7. Have measurable lesion by RECIST 1.1 criteria.
8. Karnofsky Performance Status (KPS) ≥60.
9. Patients must be willing to enroll the clinical study, and comply with the study and follow-up procedures.
10. Adequate organ and bone marrow functions:

    1. White Blood Count (WBC) ≥ 3,000/mm3 (3.0×109/L);
    2. Neutrophils≥ 1,000/mm3 (1.0×109/L);
    3. Platelets (PLT) ≥ 80,000/mm3 (80×109/L);
    4. Hemoglobin（Hb）≥ 9 g/dL (90g/L);
    5. Serum creatinine ≤ 1.5x the upper limit of normal (ULN) or creatinine clearance (CrCl)≥ 40 mL/min;
    6. Bilirubin≤ 1.5x ULN;
    7. Aspartate Aminotransferase (AST) ≤ 2.5x ULN or Alanine Aminotransferase (ALT) ≤ 2.5x ULN; patients with liver metastasis must be ≤5x ULN;
    8. International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
    9. Urine protein < 2 +; if urinary protein ≥ 2 +, the 24-hour urine protein quantification must be ≤ 1g.

Exclusion Criteria:

1. Other diseases that may have influence on this study ( such as active infection, symptomatic myocardial infarction, angina pectoris, arrhythmia, etc.).
2. Patients who received systemic anti-tumor therapy and local treatment (radiotherapy, ablation and embolization) for gastric cancer within 1 month.
3. Patients who have active autoimmune diseases and need systemic immunosuppressive therapy.
4. Life expectancy < 6 months.
5. Patients with organ allografts.
6. Women who are pregnant or nursing/breastfeeding
7. Allergic to allogeneic protein.
8. Human immunodeficiency virus (HIV) infection, untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 500 IU / ml; hepatitis C, defined as HCV-RNA higher than the detection limit of the analytical method).
9. For any other reasons, the patients are believed not suitable for participation in this study by investigators .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 6 months
  The proportion of patients with complete response(CR) or partial response(PR) as measured by RECIST 1.1 criteria.
Disease Control Rate (DCR) (PR+CR+SD) | 6 months
  The proportion of patients with complete response (CR), partial response (PR), or stable disease (SD).
Progression-free Survival (PFS) | 6 months
  The length of time during and after the treatment, that a patient lives with the disease but it does not get worse.
Health-related quality of life (QoL): 36-Item Short Form (SF-36) | 6 months
  Medical Outcomes Study 36-Item Short Form (SF-36)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (PR+CR) | 12 months
  The proportion of patients with complete response(CR) or partial response(PR) as measured by RECIST 1.1 criteria.
Disease Control Rate (DCR) (PR+CR+SD) | 12 months
  The proportion of patients with complete response (CR), partial response (PR), or stable disease (SD).
Progression-free Survival (PFS) | 12 months
  The length of time during and after the treatment, that a patient lives with the disease but it does not get worse.
Health-related quality of life (QoL): 36-Item Short Form (SF-36) | 12 months
  Medical Outcomes Study 36-Item Short Form (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Hospital of Shandong University, Jinan, Shandong, China